CLINICAL TRIAL: NCT01143909
Title: Transfusion of Fresh Frozen Plasma in Non-bleeding ICU Patients
Brief Title: Transfusion of Fresh Frozen Plasma in Non-bleeding Intensive Care Unit (ICU) Patients
Acronym: TOPIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: N.P. Juffermans, MD, PhD, Academic Medical Centre - University of Amsterdam
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ZonMw-80823109710069; NTR2262 (Registry Identifier: Dutch Trial Register)
Record Dates: First submitted 2010-06-14; First posted 2010-06-15 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2010-06

CONDITIONS: Blood Coagulation Disorders; Hemorrhage
Keywords: Fresh frozen plasma; Coagulopathy; Intensive care; Adverse effects; Lung injury
MeSH Terms: conditions — Blood Coagulation Disorders; Hemorrhage; Hemostatic Disorders; Lung Injury

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No FFP transfusion prior to intervention (Experimental): Patients with a coagulopathy (INR 1,5-3,0), who are randomized to omitting transfusion of fresh frozen plasma before they undergo an intervention.
  Interventions: Other: omitting FFP transfusion before an intervention
- FFP transfusion prior to intervention (No Intervention): Patients with a coagulopathy (INR 1,5-3,0), who are randomized to transfusion of fresh frozen plasma before they undergo an intervention. This is considered standard care.

INTERVENTIONS:
Other: omitting FFP transfusion before an intervention — In the interventional group FFP transfusion is omitted before performing a procedure (e.g. placement of central venous catheter, tracheostomy, chest tube)
  Arms: No FFP transfusion prior to intervention

SUMMARY:
With the aim to restrict inappropriate fresh frozen plasma (FFP) transfusions to critically ill patients, a randomized clinical trial will be conducted in a subgroup of intensive care (ICU) patients undergoing an invasive procedure. The objective is to assess the effectiveness and costs of omitting prophylactic FFP transfusion compared to current practice of prophylactic transfusion, in non-bleeding ICU patients with a coagulopathy.

DETAILED DESCRIPTION:
Rationale: Fresh frozen plasma (FFP) is an effective therapy to correct for a deficiency of multiple coagulation factors during bleeding. In past years, use of FFP has increased, in particular in patients on the Intensive Care Unit (ICU), and has expanded to include prophylactic use in patients with a coagulopathy prior to undergoing an invasive procedure. Retrospective studies suggest that prophylactic use of FFP does not prevent bleeding, but carries the risk of transfusion-related morbidity. However, up to 50% of FFP is administered to non-bleeding ICU patients.

Objective: With the aim to restrict inappropriate FFP transfusions to critically ill patients, a randomized clinical trial will be conducted in a subgroup of ICU patients with a coagulopathy undergoing an invasive procedure. The objective is to assess the effectiveness and costs of prophylactic FFP transfusion (current practice) compared to no prophylactic transfusion, in non-bleeding ICU patients with a coagulopathy, prior to undergoing an invasive procedure (e.g. placement of central venous catheter, tracheostomy, chest tube).

Study design: Prospective, multicentre, randomized, open-label, blinded end point evaluation (PROBE) design.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* INR >1.5 and <3.0
* undergoing invasive procedure (insertion of a central venous catheter, a chest drain, percutaneous tracheostomy)

Exclusion Criteria:

* clinically overt bleeding at the time of the procedure (excludes minor epistaxis, minor gum bleeding, microscopic hematuria, superficial bruises, or normal menses)
* thrombocytopenia of < 30 x 109/L.
* use of abciximab, tirofiban, ticlopidine or activated protein C
* use of heparin < 1 hour prior to the procedure, or low molecular weight heparin in therapeutic doses < 12 hours prior to procedure
* history of congenital or acquired coagulation factor deficiency or bleeding diathesis
* no informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2010-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Procedure-related relevant bleeding, occurring within 24 hours after the procedure. | 24 hours after the procedure
  Relevant bleeding will be defined using a validated tool for assessment of bleeding in the critically ill.
  An assessment of bleeding will be standardized and performed by an independent research physician or intensivist blinded to the transfusion strategy 1 and 24 hours after the procedure and when clinically indicated.

SECONDARY OUTCOMES:
minor bleeding within 24 hours | within 24 hours of the procedure
onset of acute lung injury within 48 hours. | 48 hours within the intervention
  Lung injury will be evaluated by P/F ratio, change in ventilator settings, chest x-ray and Lung Injury Score.
effect of FFP transfusion on coagulation parameters | within 24 hours of transfusion of FFP
  a range of coagulation parameters will be evaluated to assess efficacy of FFP transfusion in these patients
evaluation of costs | up to 28 days after inclusion
  Evaluation of costs in the two different groups will be made. Length of stay, number of ventilation days, differences in medication use, all will be taken into account.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole P Juffermans, MD, PhD, Principal Investigator — Academic Medical Centre - University of Amsterdam
Locations (4):
- Netherlands (4):
  - Diakonessenhuis, Utrecht, Utrecht
  - Academic Medical Centre - University of Amsterdam, Amsterdam
  - Ter Gooi Ziekenhuizen, Hilversum
  - Leids Universitair Medisch Centrum, Leiden

REFERENCES:
- [Derived] Straat M, Muller MC, Meijers JC, Arbous MS, Spoelstra-de Man AM, Beurskens CJ, Vroom MB, Juffermans NP. Effect of transfusion of fresh frozen plasma on parameters of endothelial condition and inflammatory status in non-bleeding critically ill patients: a prospective substudy of a randomized trial. Crit Care. 2015 Apr 15;19(1):163. doi: 10.1186/s13054-015-0828-6. PMID 25880761
- [Derived] Muller MC, Straat M, Meijers JC, Klinkspoor JH, de Jonge E, Arbous MS, Schultz MJ, Vroom MB, Juffermans NP. Fresh frozen plasma transfusion fails to influence the hemostatic balance in critically ill patients with a coagulopathy. J Thromb Haemost. 2015 Jun;13(6):989-97. doi: 10.1111/jth.12908. Epub 2015 Apr 18. PMID 25809519
- [Derived] Muller MC, de Jonge E, Arbous MS, Spoelstra-de Man AM, Karakus A, Vroom MB, Juffermans NP. Transfusion of fresh frozen plasma in non-bleeding ICU patients--TOPIC trial: study protocol for a randomized controlled trial. Trials. 2011 Dec 23;12:266. doi: 10.1186/1745-6215-12-266. PMID 22196464